CLINICAL TRIAL: NCT00454545
Title: Atorvastatin in Moderate Active Crohns Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Skane University Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 010-02
Record Dates: First submitted 2007-03-29; First posted 2007-03-30 (Estimated); Last update posted 2007-10-22 (Estimated); Status verified 2007-10

CONDITIONS: Crohns Disease
MeSH Terms: conditions — Crohn Disease | interventions — Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Atorvastatin

SUMMARY:
Open pilot study to collect information regarding the effect of atorvastatin on patients with active Crohns disease.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Crohns disease
* C-reactive protein level > 2 mg/L in absence of an infection
* Fecal calprotectin > 250 mg/kg or CDAI > 150

Exclusion Criteria:

* CDAI > 450
* Prednisolone dosage above 15 mg/day

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2006-10; Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Inflammatory markers in plasma before and after treatment.

SECONDARY OUTCOMES:
Change in clinical activity index and mucosal inflammation after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Olof Grip, MD, PhD, Principal Investigator — Malmo University Hospital, Region Skåne; Anders Bredberg, MD, PhD, Study Chair — Malmo University Hospital, Region Skåne; Gunnel Bredberg, MD, PhD, Study Chair — Malmo University Hospital, Region Skåne
Locations (1):
- Department of Medicine, Division of Gastroenterology and Hepatology, Malmo, Sweden

REFERENCES:
- [Derived] Grip O, Janciauskiene S. Atorvastatin reduces plasma levels of chemokine (CXCL10) in patients with Crohn's disease. PLoS One. 2009;4(5):e5263. doi: 10.1371/journal.pone.0005263. Epub 2009 May 6. PMID 19421322